CLINICAL TRIAL: NCT00912574
Title: Evaluation of the Effects of Local GM-CSF-in-Adjuvant Administration on Dendritic Cells in Skin of Melanoma Patients and in Sentinel Lymph Nodes
Brief Title: Evaluation of the Effects of Local Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Adjuvant Administration on Dendritic Cells in Skin of Melanoma Patients and in Sentinel Lymph Nodes: MEL38
Acronym: MEL38
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Craig L Slingluff MD, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8380
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Melanoma
Keywords: Melanoma; adjuvant; dendritic cells; vaccine
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; Granulocyte-Macrophage Colony-Stimulating Factor; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline (Active Comparator): first of 4 arms: injection: 1 ml saline
  Interventions: Drug: Saline
- GM-CSF (Active Comparator): Second of 4 arms: injection: specified dose of GM-CSF in 1 ml saline
  Interventions: Drug: GM-CSF-in-adjuvant
- 0.5 ml Montanide ISA-51 adjuvant and 0.5 ml saline (Active Comparator): Third of 4 arms: injection: 0.5 ml Montanide ISA-51 adjuvant and 0.5 ml saline
  Interventions: Drug: Montanide ISA-51
- GM-CSF in 0.5 ml slaine plus 0.5 ml Montanide ISA-51 adjuvant (Active Comparator): Fourth of 4 arms: injection: specified dose of GM-CSF in 0.5 ml slaine plus 0.5 ml Montanide ISA-51 adjuvant
  Interventions: Biological: GM-CSF and Montanide ISA-51

INTERVENTIONS:
Drug: GM-CSF-in-adjuvant — For each injection, patients will receive the following: In stage 1: Patients will be injected with a 1 ml emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant, in skin adjacent to a melanoma biopsy scar.
  In stage 2: Patients will be randomized to receive an injection of one of the following in skin adjacent to the melanoma biopsy scar at one of two time points:
  1. 1 ml saline
  2. specified dose of GM-CSF in 1 ml saline
  3. an emulsion of 0.5ml Montanide ISA-51 adjuvant and 0.5 ml saline
  4. an emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant
  Arms: GM-CSF
Drug: Montanide ISA-51 — For each injection, patients will receive the following: In stage 1: Patients will be injected with a 1 ml emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant, in skin adjacent to a melanoma biopsy scar.
  In stage 2: Patients will be randomized to receive an injection of one of the following in skin adjacent to the melanoma biopsy scar at one of two time points:
  1. 1 ml saline
  2. specified dose of GM-CSF in 1 ml saline
  3. an emulsion of 0.5ml Montanide ISA-51 adjuvant and 0.5 ml saline
  4. an emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant
  Arms: 0.5 ml Montanide ISA-51 adjuvant and 0.5 ml saline
Biological: GM-CSF and Montanide ISA-51 — For each injection, patients will receive the following: In stage 1: Patients will be injected with a 1 ml emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant, in skin adjacent to a melanoma biopsy scar.
  In stage 2: Patients will be randomized to receive an injection of one of the following in skin adjacent to the melanoma biopsy scar at one of two time points:
  1. 1 ml saline
  2. specified dose of GM-CSF in 1 ml saline
  3. an emulsion of 0.5ml Montanide ISA-51 adjuvant and 0.5 ml saline
  4. an emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant
  Arms: GM-CSF in 0.5 ml slaine plus 0.5 ml Montanide ISA-51 adjuvant
Drug: Saline — For each injection, patients will receive the following: In stage 1: Patients will be injected with a 1 ml emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant, in skin adjacent to a melanoma biopsy scar.
  In stage 2: Patients will be randomized to receive an injection of one of the following in skin adjacent to the melanoma biopsy scar at one of two time points:
  1. 1 ml saline
  2. specified dose of GM-CSF in 1 ml saline
  3. an emulsion of 0.5ml Montanide ISA-51 adjuvant and 0.5 ml saline
  4. an emulsion of specified dose of GM-CSF in 0.5 ml saline plus 0.5 ml Montanide ISA-51 adjuvant
  Arms: Saline

SUMMARY:
Goal: To characterize the cellular events that occur in vivo after vaccination with an emulsion of GMCSF-in-adjuvant.

Design: Open-label, single dose study in two stages.

DETAILED DESCRIPTION:
Regimen: Each injection will be administered to patients with clinical stage I or II melanoma, who have had complete excision of a primary melanoma, but prior to wide excision with or without sentinel node biopsy as definitive surgical therapy.

In Stage 1: Patients will be injected with a 1 ml emulsion containing GM-CSF in saline plus Montanide ISA-51 adjuvant, in skin adjacent to a melanoma biopsy scar.

In Stage 2: Patients will be randomized to receive an injection of one of the following in skin adjacent to the melanoma biopsy scar:

1. 1 ml saline
2. GM-CSF in 1 ml saline
3. an emulsion of Montanide ISA-51 adjuvant and saline
4. an emulsion of GM-CSF in saline plus ml Montanide ISA-51 adjuvant. All vaccines will be administered intradermally. After the injection, each patient will undergo wide excision of the melanoma site, with or without sentinel node biopsy, as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed, by histologic and clinical examination, with resected AJCC stage I or II melanoma.
* Patients who have any evidence of metastasis will not be eligible.
* All patients must have:

  1. Karnofsky performance of 80% or higher
  2. ECOG performance status of 0 or 1
  3. Ability and willingness to give informed consent
* Laboratory parameters as follows:

  1. ANC: 90% of lower limit of normal (LLN) to 120% of upper limit of normal (ULN)
  2. Platelets: 100-500 x 103/uL
  3. Hgb: 90% LLN to 120% ULN
  4. Hepatic:

     1. AST, ALT, Bilirubin, and Alk phos within normal limits,
     2. LDH up to 1.2 x ULN
  5. Renal:

     1. Creatinine up to 1.5 x ULN
* Age 18-85 years at the time of study entry.

Exclusion Criteria:

* Patients who are currently receiving cytotoxic chemotherapy, interferon, or radiation or who have received this therapy within the preceding 12 weeks.
* Patients with known or suspected allergies to any component of the vaccine.
* Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded:

  * Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents),
  * Allergy desensitization injections,
  * Corticosteroids, administered parenterally or orally. Topical corticosteroids are acceptable.
  * Any growth factors, Interleukin-2 or other interleukins.
* Pregnancy or the possibility of becoming pregnant during vaccine administration. Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the injection.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified according to the New York Heart Association classification as having Class III or IV heart disease.
* Patients with serious symptomatic active pulmonary disease, with pleural effusions, or with a history of pulmonary edema.
* Patients who have systemic autoimmune disease with visceral involvement.
* Patients with clinically apparent skin infection or other clinically evident inflammation involving the skin adjacent to the melanoma biopsy scar.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number of dendritic cells (total and mature) accumulating in the dermis after administration of the adjuvant
Proportion of the sentinel node occupied by dendritic cells (total and mature)

SECONDARY OUTCOMES:
Time to maximal dendritic cell infiltration into the dermis

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States